# The Effects of Yi Jin Bang Exercise on Shoulder Health of Adults

Date: 12/19/2021

#### Information sheet and Consent form

Prof. HUI, Stanley Sai-chuen, Professor in the Department of Sports Science and Physical Education in The Chinese University of Hong Kong, will conduct a project entitled "The Effects of Yi Jin Bang Exercise on Shoulder Health of Adults". You are sincerely invited to participate in this study.

#### INFORMATION

The purpose of this study is to examine the effects of Yi Jin Bang exercise on shoulder health of adults. Hong Kong Chinese adults with subacromial pain syndrome, aged 18-65 years old will be recruited in this study. You will be randomly assigned into one of the following three groups: group 1: Yi Jin Bang, group 2: usual exercise therapy, or group 3: waitlist control group. All three groups will receive relevant fitness tests, three times during the period of 10 weeks, including pain intensity test, functional disability test, flexibility test, and muscular endurance test at the Fitness Laboratory of the Department of Sports Science and Physical Education, The Chinese University of Hong Kong. Participants in groups 1 & 2 will be invited to attend three tutorial sessions immediately after the initial fitness tests, where participants can learn the Yi Jin Bang exercise or the usual exercise therapy under the guidance of instructors, followed by a 10-week exercise training. Participants in group 3 will attend the same tutorial sessions after 10 weeks, then will be provided exercise training in the next 10 weeks. In addition, participants in all three groups should come to the Fitness Laboratory to attend the first exercise session.

#### The details of each group include:

Group 1: The Yi Jin Bang group. Participants in group 1 will engage in initial fitness assessment, follow by 10 weeks of home-based Yi Jin Bang exercise training [four times a week, which consists of 10 minutes of warm-up, 18 minutes of Yi Jin Bang (10 movements), and 10 minutes of cool-down]. Additionally, after the first exercise session, the second fitness assessment will be provided. After 10 weeks, the third fitness assessment will be provided.

Group 2: The usual exercise therapy group. Participants in group 2 will engage in initial fitness assessment, follow by 10 weeks of standardized home-based stretching and strengthening exercise program. This program includes four stretching exercises and seven resistance-strengthening exercises and will be performed four times per week. Additionally, after the first exercise session, the second fitness assessment will be provided. After 10 weeks, the third fitness assessment will be provided.

Group 3: The waitlist control group. Participants in group 3 will also attend the first exercise session. Participants will be instructed to watch an educational video about shoulder pain during the session. Participants will engage in fitness assessment at the beginning (week 1), after the first exercise session, and at week 10. Then participants will be provided a 10 weeks either Yi Jin Bang or usual exercise therapy training.

## **BENEFITS**

You will better understand the condition of your affected shoulder and may obtain corresponding treatment effects. In addition, you will receive a supermarket voucher worth HKD \$200 when you finish the tests, including the waitlist control group. You will not be charged for the study article/service.

# FORESEEABLE RISKS

There is no reasonably foreseeable risk or discomfort in this study. To ensure the safety, the study protocol stated that if the participant cannot complete the physical activity at any intensity level, he/she will be terminated from the test, and will not be proceeded to the next intensity level. Furthermore, preparticipation health screening (PAR-Q) will be conducted according to American College of Sports Medicine (ACSM) guidelines for all participants in order to minimize the risks.

## **CONFIDENTIALITY**

All the data record sheets of participants will be filed with a specific code number. All the files will be kept by the principle investigator and classified as confidential. The results of the tests of all subjects will be reported in aggregate terms and individual responses will not be disclosed. The subjects' personal particulars will not be recorded in data file other than the participant's code. All data files will be stored with security codes. All data files and data sheets will be destroyed three years after the completion of the research study.

#### **ENQUIRY:**

If you have questions at any time about the study or the procedures, you may contact the Principal Investigator: Prof. Stanley Sai-chuen HUI (Tel: 3943 6081; Email: hui2162@cuhk.edu.hk) or Research Assistant: Mr. Jinde Liu (Tel: 3943 5253; Email: jinde.liu@link.cuhk.edu.hk). If you have any questions about the study and the research staffs, you can also contact Join CUHK-NTEC Clinical Research Ethics Committee (Tel: 3505 3935; email: crec@cuhk.edu.hk). Due to this study approved by Join CUHK-NTEC Clinical Research Ethics Committee, they have the legal right to see the participants' information for proceeding the ethical approval.

# **SCOPE of CONSENT:**

Your participation in this study is voluntary, you may decline to participate without penalty. If you decide to participate, you may withdraw from the study at any time without penalty and without loss of benefits to which you are otherwise entitled. If you withdraw from the study your data will be destroyed.

| <b>Declaration:</b> I have read this form and understoassigned into group | | ood the purpose as well as the measurement items. I am being randomly, and agree to voluntarily take part in the study. | | |
|---|---|---|---|---|
| I acknowledge that without negative co | _ | ht to question any part | t of the procedure a | nd can withdraw at any time |
| Witness | Name: | Witness's | Signature: | Date: |
| Participant | Name: | Participant's | Signature: | Date: |
| Investigator | Name: | Investigator's | Signature: | Date: |